CLINICAL TRIAL: NCT07083765
Title: A Prospective Multicenter, Blinded, Sham Procedure-Controlled Trial of Renal Denervation Using the Dehydrated Alcohol Injection, USP Administered With the Peregrine System™ Infusion Catheter in Subjects With Hypertension, in the Absence of Antihypertensive Medications
Brief Title: Renal Artery Denervation Assessment Without Antihypertensive Medication Regimen (RADAR)
Acronym: RADAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ablative Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR0041
Record Dates: First submitted 2025-05-12; First posted 2025-07-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Hypertension,Essential
Keywords: Renal denervation; Neurolysis
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Treatment arm: renal denervation performed with dehydrated alcohol injection, USP administered via the Peregrine System™ Infusion Catheter.
  Sham Control Arm: only renal angiography performed
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Renal denervation performed with dehydrated alcohol injection, USP administered via the Peregrine System™ Infusion Catheter.
  Interventions: Drug: Dehydrated Alcohol Injection, USP
- Sham Control Arm (Sham Comparator): Only renal angiography performed
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Drug: Dehydrated Alcohol Injection, USP — Alcohol is directly infused/delivered to the adventitial and periadventitial space of the renal arteries
  Other Names: Alcohol
  Arms: Treatment Arm
Procedure: Sham procedure — Endovascular, renal angiography
  Arms: Sham Control Arm

SUMMARY:
To obtain an assessment of the efficacy and safety of renal denervation by dehydrated alcohol injection, USP administered via the Peregrine System™ Infusion Catheter in hypertensive subjects in the absence of antihypertensive medications.

DETAILED DESCRIPTION:
This Phase 3, prospective, randomized, blinded, sham procedure-controlled, multicenter study will assess the efficacy and safety of renal denervation by alcohol-mediated neurolysis using the Peregrine Catheter in hypertensive subjects in the absence of antihypertensive medications. Subjects with a documented history of uncontrolled hypertension who are taking 0, 1, or 2 antihypertensive medications at enrollment will be recruited. After providing written informed consent, subjects will undergo screening assessments to assess eligibility for the study. Eligible subjects will then enter a run in period during which they will take no antihypertensive medications. Subjects who continue to be eligible at the end of the run-in period will complete the study Baseline visit and remain without taking antihypertensive medications. Subjects who continue to be eligible after the completion of the Baseline visit will attend the study site and will be randomized to either the Treatment Arm (renal denervation using the Peregrine Catheter) or the Sham Control Arm (renal angiography only).

After study unblinding, crossover from the Sham Control Arm to the Treatment Arm may be allowed, at the discretion of the treating investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Has 2 office blood pressure measurements with a mean office systolic blood pressure (SBP) of ≥150 mmHg and ≤180 mmHg, AND a mean office diastolic blood pressure (DBP) of ≥90 mmHg.
2. Documented history of uncontrolled hypertension and is currently taking 1 or 2 antihypertensive medications.
3. Is willing to discontinue any current antihypertensive medications for at least 13 weeks (5-week pre-procedure and 8-week post-procedure).
4. Has a mean 24-hour ambulatory SBP of ≥140 mmHg and ≤170 mmHg with required valid readings.

Exclusion Criteria:

1. Has renal artery anatomy abnormalities.
2. Has previously undergone renal denervation.
3. Has an estimated glomerular filtration rate (eGFR) of ≤45 mL/min/1.73 m2, based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation; or is on chronic renal replacement therapy.
4. Has documented untreated sleep apnea.
5. Has any of the following conditions: severe cardiac valve stenosis, heart failure (New York Heart Association [NYHA] Class III or IV), chronic atrial fibrillation (defined as at least one documented episode in the 12 months before study entry), and known primary pulmonary hypertension (>60 mmHg pulmonary artery or right ventricular systolic pressure).
6. Is pregnant or lactating at the time of enrollment or planning to become pregnant during the trial time period (female subjects only).
7. Is being treated chronically (e.g. daily use) with NSAIDs, immunosuppressive medications, or immunosuppressive doses of steroids. Aspirin therapy and nasal pulmonary inhalants are allowed.
8. Has a history of myocardial infarction, unstable angina pectoris, or stroke/TIA within 6 months prior to the planned procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Systolic Ambulatory Blood Pressure at 8 weeks | Baseline to 8 weeks post-treatment
  Change from baseline in mean 24-hour ambulatory systolic blood pressure

SECONDARY OUTCOMES:
Change in Office SBP at 8 Weeks | Baseline to 8 weeks post-treatment
  Change from Baseline in mean office SBP to Week 8
Change in Office DBP at 8 Weeks | Baseline to 8 weeks post-treatment
  Change from Baseline in mean office DBP to Week 8
Changes in Diastolic Ambulatory Blood Pressure at 8 Weeks | Baseline to 8 weeks post-treatment
  Change from baseline in mean 24-hour ambulatory diastolic blood pressure at 8 weeks post-procedure
Changes in Systolic Ambulatory Blood Pressure at 6 Months | Baseline to 6 months post-treatment
  Change from baseline in mean 24-hour ambulatory systolic blood pressure at 6 months post-procedure
Changes in Diastolic Ambulatory Blood Pressure at 6 Months | Baseline to 6 months post-treatment
  Change from baseline in mean 24-hour ambulatory diastolic blood pressure at 6 months post-procedure
Changes in Mean Daytime Ambulatory SBP at 8 Weeks | Baseline to 8 weeks post-treatment
  Change from baseline in mean daytime systolic blood pressure at 8 weeks post-procedure
Changes in Mean Daytime Ambulatory SBP at 6 Months | Baseline to 6 months post-treatment
  Change from baseline in mean daytime systolic blood pressure at 6 months post-procedure
Changes in Mean Daytime Ambulatory DBP at 8 Weeks | Baseline to 8 weeks post-treatment
  Change from baseline in mean daytime diastolic blood pressure at 8 weeks post-procedure
Changes in Mean Daytime Ambulatory DBP at 6 Months | Baseline to 6 months post-treatment
  Change from baseline in mean daytime diastolic blood pressure at 6 months post-procedure
Changes in Mean Nighttime Ambulatory SBP at 8 Weeks | Baseline to 8 weeks post-treatment
  Change from baseline in mean nighttime systolic blood pressure at 8 weeks post-procedure
Changes in Mean Nighttime Ambulatory SBP at 6 Months | Baseline to 6 months post-treatment
  Change from baseline in mean nighttime systolic blood pressure at 6 months post-procedure
Changes in Mean Nighttime Ambulatory DBP at 8 Weeks | Baseline to 8 weeks post-treatment
  Change from baseline in mean nighttime diastolic blood pressure at 8 weeks post-procedure
Changes in Mean Nighttime Ambulatory DBP at 6 Months | Baseline to 6 months post-treatment
  Change from baseline in mean nighttime diastolic blood pressure at 6 months post-procedure
Change in Office SBP at 6 Months | Baseline to 6 months post-treatment
  Change from Baseline in mean office DBP at 6 months post-procedure
Change in Office DBP at 6 Months | Baseline to 6 months post-treatment
  Change from Baseline in mean office DBP to Week 8 at 6 months post-procedure
Use of Antihypertensive Medication(s) at 8 Weeks | 8 weeks post-treatment
  Use of antihypertensive medication at 8 weeks post-procedure
Use of antihypertensive medication(s) from 8 Weeks to 6 Months | 6 months post-treatment
  Change in use of antihypertensive medication(s) from 8 Weeks to 6 Months post procedure (titrated according to standardized formula to maintain a target SBP of <140 mmHg and ≥90 mmHg)
Number of Participants With Major Adverse Events (MAEs) | 30 days post-treatment
  Number of participants with major adverse events (MAEs) 30 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weber, MD, Principal Investigator — SUNY Downstate Medical Center and College of Medicine; David Kandzari, MD, Principal Investigator — Piedmont Healthcare; Felix Mahfoud, Prof.Dr. med, Principal Investigator — University of Basel; Atul Pathak, Prof., Principal Investigator — Princess Grace Hospital, Monaco
Locations (1):
- Tennova Turkey Creek Medical Center, Knoxville, Tennessee, United States